CLINICAL TRIAL: NCT04614701
Title: Correlation of Carotid Flow Time and Cardiac Output With Preload Augmentation in Patients With COVID-19.
Brief Title: Correlation of Carotid Flow Time and Cardiac Output.
Status: Withdrawn | Type: Observational
Why Stopped: The co and principal investigator, due to limited resources and timing, have decided to withdrawal the study and close.
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rakesh C. Arora, Section Head Cardiac Surgery, St. Boniface Hospital
Other Study IDs: HS24296
Record Dates: First submitted 2020-10-21; First posted 2020-11-04 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Volume Responsiveness
Keywords: volume responsiveness, ultrasound, fluid responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Carotid Artery Ultrasound Measure — Cardiac output will be assessed by measuring the LVOT diameter in parasternal long-axis window and the LVOT VTI in apical-four window. Carotid artery flow will be measured on the right neck 1-2cm from the bifurcation of the common carotid artery. All measurements will be taken with participants supine and the head of the bed elevated to 45°. measures all at 3 minute intervals.
  1. One-leg compression test: Thigh-sized blood pressure cuff inflated to 60mmHg on middle part of one thigh for 60 seconds. LVOT and CCA measurements taken separately.
  2. Two-leg compression test: Thigh-sized blood pressure cuff inflated on middle part of both thighs for 60 seconds. LVOT and CCA measurements taken separately.
  3. Passive leg raise test: Bed adjusted to place participant at 0° and legs elevated at 45° by use of pillows. After 1 minute, measurements repeated. LVOT and CCA measurements taken separately.

SUMMARY:
Assessment of common carotid artery flow is more easily done and can be taught more broadly than transthoracic echocardiography, providing a greater number of clinicians a tool to assess volume responsiveness. These assessments are of great importance to patients with COVID-19, who often present with hypotension requiring fluids, which must be balanced against limiting fluid administration to minimize pulmonary edema.

DETAILED DESCRIPTION:
Optimizing volume status for patients in shock is of critical importance to their outcomes, both in the provision of helpful, and avoidance of harmful fluid volumes. As such, much work has been done to develop and assess measures of volume responsiveness; that is, tests that indicate whether additional fluid administration will increase cardiac output by at least 10%. The passive leg raise (PLR) providing a reversible "auto-bolus" has been demonstrated to be the most predictive assessment of fluid responsiveness.

Recent studies of changes in carotid artery blood flow suggest it can be used as a surrogate for changes in cardiac output with moderate reliability. This has been assessed in several populations with anticipated changes in volume status (e.g. before/after blood donation), and more recently assessed by Sidor et al. against several preload augmenting maneuvers. Interestingly, while decreasing preload resulted in a decrease in cardiac output and systolic carotid blood flow, it did not result in a decrease in corrected carotid flow time, although a PLR produced an expected increase in all measures.

In our study we seek to validate these results, questioning if there is a lower limit of corrected carotid flow time that de-couples the relationship between carotid systolic flow and corrected carotid flow time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to hospital with diagnosed COVID-19, on up to 6L oxygen, and able to undergo leg compression testing and passive leg raise.

Exclusion Criteria:

* known cardiac disease, carotid atherosclerosis, prior right-sided neck surgery, chest wall deformity, or deep-venous thrombosis identified on admission

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 20 adult (age 18-80) patients admitted to the hospital with COVID-19 requiring supplemental oxygen, up to 6L, willing to undergo transthoracic and right carotid ultrasonography.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in measured LVOT VTI by bedside echocardiography | Through study completion, up to 1 year
  Measurements for this parameter will be obtained at baseline, following one-leg and two-leg compression tests, and following passive leg raise
Changed in corrected carotid artery flow time as measured by bedside carotid artery ultrasonography. | Through study completion, up to 1 year
  Measurements for this parameter will be obtained at baseline, following one-leg and two-leg compression tests, and following passive leg raise.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh C Arora, MD, Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No